CLINICAL TRIAL: NCT00415675
Title: Assessing the Magnitude and Potential Impact of Respiration-Induced Three-Dimensional Motion of Tumors and Normal Tissues Using Four-Dimensional CT Technology
Brief Title: Respiratory Tumor and Normal Tissue Motion
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2003-0962
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Lung Cancer; Abdominal Cancer
Keywords: Lung Cancer; Abdominal Cancer; Tissue Motion; Breathing; Motion CT Scans
MeSH Terms: conditions — Lung Neoplasms; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Respiratory Tumor + Normal Tissue Motion
  Interventions: Procedure: Motion CT Scans

INTERVENTIONS:
Procedure: Motion CT Scans — A total of up to 12 scanning sessions used to understand how the tumor and other organs move while breathing.

SUMMARY:
Primary Objectives:

* To collect accurate and reliable respiration-induced anatomic structure motion data using four-dimensional (4-D) imaging technology.
* To analyze these data to study respiration-induced variations and patterns in variations of positions, shapes and volumes of tumors and normal anatomic structures in the thorax and abdomen over a breathing cycle, from one breathing cycle to the next, day-to-day and over the course of radiotherapy.
* To assess dosimetric and potential clinical consequences of respiratory motion in the current practice of radiotherapy through preclinical treatment simulation (treatment planning) studies.
* To quantify the potential consequences of explicitly accounting for respiration-induced motion on dose distributions and outcome (tumor control probabilities and normal tissue complication probabilities) through preclinical treatment simulation studies.

Secondary Objectives:

* To investigate the feasibility of using patient training to regulate patient breathing and improve the quality of images and to stratify patients for their eligibility for respiratory-correlated imaging and radiotherapy and for the implementation of various strategies for mitigation of respiratory-induced motion.
* To assess the degree of correlation of the marker (or internal anatomic structure such as diaphragm) being tracked as surrogate of breathing with the motion of structures and the intra-fraction and inter-fraction reproducibility of such correlation.
* To quantify the effects of radiation therapy on the patterns of respiratory-induced motion of structures through preclinical treatment simulation studies.
* To compare various strategies for either accounting for or mitigating respiration-induced motion in the planning and delivery of radiation therapy.

DETAILED DESCRIPTION:
You will be taking part in this study while you receive radiotherapy treatment for your tumor.

You will be trained to breathe in a certain way that will help the study staff to perform motion CT scans. You may be asked to breathe normally, or hold your breath, or breathe while following a TV monitor. On the monitor, you will be viewing your breathing trace and using the trace to regulate your breathing as instructed by the health professionals.

While you are in the right position for the scan, the study staff will perform motion CT scans. A total of up to 12 scanning sessions will be held over your entire course of radiotherapy. The first scanning session may last from 45 to 90 minutes, but later sessions may be shorter. These CT scans are separate from the routine CT scans you may receive as part of regular radiation treatment planning.

Scans may be taken at various periods of time. The scans can be taken one right after another, or with a short separation between them. One scan can be taken on the first day, and the next scan on the next day, or up to a week later.

By looking at the scans, researchers can better understand how your tumor and other organs move from breath to breath, from day to day, and from week to week.

This is an investigational study. About 210 patients with the same tumor location as you will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathological diagnosis of cancer in the thorax or abdomen.
2. Patients must be planned to have radiation therapy delivered over at least 4 weeks (a minimum standard duration of curative radiotherapy).
3. Patients must be able to lie flat for the duration of the CT image acquisition sessions.

Exclusion Criteria:

1. Patients who are neither able to breathe nor hold breath in a regular and reproducible manner will be removed from the study as being ineligible. Breathing or breath-holding regularity determination will be based on respiration traces acquired with the RPM system.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants with Abdominal or Lung Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2004-11; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Indices of Respiration-induced Anatomic Structure Motion, Structure Volume + Structure Shape Changes | 3 Years Data Collection: Up to 12 scanning sessions per patient from baseline to completion of radiotherapy (minimally 4 week treatment)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Cox, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org